CLINICAL TRIAL: NCT04942795
Title: se of ADAPT Assisted by a Compliant Balloon (ADAPT-AB) When ADAPT Fails for Acute Stroke Thrombectomy
Brief Title: Use of a Compliant Balloon for Large Bore Catheter Navigation in Mechanical Thrombectomy for Stroke: a Retrospective Study
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 21Imagerie01
Record Dates: First submitted 2021-06-24; First posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Mechanical thrombectomy: Patients who underwent mechanical thrombectomy for large vessel occlusion of the anterior circulation
  Interventions: Device: Compliant balloon

INTERVENTIONS:
Device: Compliant balloon — Use of a compliant balloon when ADAPT fails to reach the clot site

SUMMARY:
The superiority of mechanical thrombectomy (MT) in patients with acute ischemic stroke from large vessel occlusion compared to standard medical therapy alone has been demonstrated by several randomized clinical trials and become the standard of care for these patients. A direct aspiration first pass technique (ADAPT) for the endovascular treatment of stroke using a large-bore catheter has been reported to be an effective method of achieving MT. Recent studies reported that ADAPT is as efficient and safe as stent retrievers, with a similar successful recanalization rate, but may have better functional outcomes, fewer procedure related-adverse events, and a tendency for faster revascularization compared to the stent-retriever thrombectomy.

However, navigation of a large-bore aspiration catheter is not always possible due to unsuccessful passage of the ophthalmic artery origin ("ledge effect") or tortuous vascular anatomy. The coaxial technique comprises guiding the large-bore catheter with a smaller inner catheter and can facilitate distal access. However, there is a gap between the inner catheter and the distal tip of the large-bore outer catheter that creates a risk of damaging the vessel wall and causing dissection or subarachnoid hemorrhage. Even with this coaxial technique, it is not always possible to reach the clot site with the large-bore catheter. To decrease the gap between the two catheters, several authors have used, in place of the inner microcatheter, a compliant balloon catheter positioned and inflated at the distal tip of the large-bore catheter. The aim of the present study was to evaluate the safety and efficacy of ADAPT assisted by a compliant balloon (ADAPT-AB) when ADAPT using the coaxial technique fails to reach the clot site.

ELIGIBILITY:
Inclusion Criteria:

* Endovascular therapy were large arterial occlusions proven by MR angiography,
* Alberta Stroke Program Early CT Score (ASPECTS) >5 on MRI,
* Baseline National Institutes of Health Stroke Scale (NIHSS) score >5.

If eligible, patients received intravenous thrombolysis (IVT).

Exclusion criteria:

- Vertebro-basilar occlusion

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent an endovascular procedure for acute stroke in a single center from November 2018 to February 2020 were included in the study
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Efficacity to reach the clot site when using an inner balloon | Day 0
  Number of patients for whom the balloon made it possible to reach the clot

SECONDARY OUTCOMES:
Clinical status at 3 month | Month 3
  Modified Rankin Score
Endovascular Complication | Day 0
  Number of dissection or vasospasm when using the balloon

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NICE, Nice, France